CLINICAL TRIAL: NCT07121387
Title: A Real-World Retrospective Cohort Analysis of SMARCA4-Deficient Advanced Lung Cancer
Brief Title: A Retrospective Cohort Analysis of SMARCA4-Deficient Lung Cancer
Status: Completed | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Yayi He, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: L23(357)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: SMARCA4-Deficient Tumor; NSCLC (Advanced Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SMARCA4-Deficient group
- SMARCA4-Intact group

SUMMARY:
This is a single-center retrospective analysis to explore the clinical characteristics, therapeutic efficacy, and tumor immune microenvironment of SMARCA4-deficient advanced non-small-cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage III-IV NSCLC according to the American Joint Committee on Cancer staging criteria (7th edition);
* Lesions are measurable according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1;
* Receiving first-line immunotherapy or chemotherapy as anti-tumor treatment.

Exclusion Criteria:

* SMARCA4 gene test was not performed;
* Not receive treatment;
* Lost to follow-up after one treatment cycle.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The clinical information of 221 patients with advanced non-small cell lung cancer from the Department of Oncology of Shanghai Pulmonary Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 5 years
  Time from the beginning of first-line therapy to the first progression (PD) in patients with lung cancer

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Overall survival (OS) is defined as the duration from the beginning of first-line therapy until death due to any cause. Subjects who are still alive at the end of the study observation period will be censored at the time of last known vital status.
Objective Response Rate (ORR) | 5 years
  The proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Disease control rate (DCR) | 5 years
  Disease control rate (DCR) was defined as the proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1).

OTHER OUTCOMES:
The correlation between tumor immune microenvironment and therapeutic efficacy | 5 years
  Multiplex immunofluorescence staining was performed on pathological specimens from individuals diagnosed with SMARCA4-deficient lung cancer who underwent immune combination chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No